CLINICAL TRIAL: NCT06431269
Title: Feasibility and Efficiency of Screening for Neurodevelopmental Disorders by an Advanced Practice Nurse in Children With Congenital Heart Disease
Acronym: NEURODEV-IPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL21_0291; ID-RCB (Registry Identifier: 2024-A00552-45)
Record Dates: First submitted 2024-05-17; First posted 2024-05-28 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-06

CONDITIONS: Congenital Heart Disease in Children; Neurodevelopmental Disorders
Keywords: congenital heart disease; neurodevelopmental screening; advanced practice nurse; organization of care; neuropsychological assessment
MeSH Terms: conditions — Neurodevelopmental Disorders; Heart Defects, Congenital | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Screening for neurodevelopmental disorders by an advanced practice nurse (Experimental)
  Interventions: Other: Screening for neurodevelopmental disorders by an advanced practice nurse

INTERVENTIONS:
Other: Screening for neurodevelopmental disorders by an advanced practice nurse — Screening for neurodevelopmental disorders by an advanced practice nurse with Ages & Stages Questionnaires (ASQ-3) and Haute Autorité de Santé (HAS) identification scale

SUMMARY:
Feasibility and efficiency of Screening for Neurodevelopmental Disorders by an Advanced Practice Nurse in Children aged 1 to 5 with Congenital Heart Disease

DETAILED DESCRIPTION:
Congenital heart disease (CHD) is the leading cause of birth defects. Over 90% of children born with CHD reach adulthood. 50% of them will develop a neurodevelopmental disorder (NDD) that could affect life and long-term prognosis, including scholar and social integration and health related quality of life.

In France, there is a lack of medical resources to screen NDD in this population and to refer patients for appropriate and early treatment.

Investigators plan to propose a systematic early screening of NDD by an Advanced Practice Nurse (APN) during the usual cardiac follow-up. Children with CHD aged 1 to 5 will be included. If NDD is suspected, the patient will be referred to a neuropsychologist for NDD diagnosis confirmation and management planning. Patients with higher NDD risks (neonatal cardiac surgery) will benefit from a systematic neuropsychologist evaluation.

This study will investigate the feasibility and performance of an APN screening in this NDD-high risk population.

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart disease with stable status defined by last operation >3 months, no cardiac decompensation in the last 3 months, no planned surgery within 6 months after the inclusion
* Cardiac surgery and/or catheter-based cardiac intervention(s) during the first year of life,
* Patient aged 1 to 5 years.
* No previous medical diagnosis of NDD
* Parental or legal guardian's consent.
* Social security affiliation (for France only)

Exclusion Criteria:

* Patients with a genetic or poly-malformative syndrome with known neurological impairment.
* Neurodevelopmental disorder already known/treated
* Neurodevelopmental status evaluation within the last 6 months.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 270 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Sensibility of the IPA screening for neurodevelopmental disorder (NDD) on the whole population studied | 4 months (to obtain the neurophysiologist assessment)
  This will be evaluated by comparing the results of the IPA screening (using both HAS scale and ASQ-3 parent's questionnaire) with results of the advanced neuropsychologist assessment. A positive IPA screening is defined by a NDD alert using the HAS scale and/or the ASQ-3 parent's questionnaire. The advanced neuropsychologist assessment will be done only for patients with CHD with a positive IPA screening.

SECONDARY OUTCOMES:
Feasibility of the IPA screening for NDD | 18 months
  This rate will be calculated by dividing the complete IPA screenings (including HAS and the ASQ-3 parent's questionnaire) and children coming to the Complex Congenital Heart Defects consultation during the study period.
Performance (sensibility) of the IPA screening for NDD on the NDD high risk population | 4 months (to obtain the neurophysiologist assessment)
  This will be evaluated by comparing the results of the IPA screening (using both HAS scale and ASQ-3 parent's questionnaire) with results of the advanced neuropsychologist assessment. A positive IPA screening is defined by a NDD alert using the HAS scale and/or the ASQ-3 parent's questionnaire. The advanced neuropsychologist assessment will be done only for patients with CHD with a positive IPA screening.
Performance (specificity) of the IPA screening for NDD on the NDD high risk population | 4 months (to obtain the neurophysiologist assessment)
  This will be evaluated by comparing the results of the IPA screening (using both HAS scale and ASQ-3 parent's questionnaire) with results of the advanced neuropsychologist assessment. A positive IPA screening is defined by a NDD alert using the HAS scale and/or the ASQ-3 parent's questionnaire. The advanced neuropsychologist assessment will be done only for patients with CHD with a positive IPA screening.
Performance (positive predictive value) of the IPA screening for NDD on the NDD high risk population | 4 months (to obtain the neurophysiologist assessment)
  This will be evaluated by comparing the results of the IPA screening (using both HAS scale and ASQ-3 parent's questionnaire) with results of the advanced neuropsychologist assessment. A positive IPA screening is defined by a NDD alert using the HAS scale and/or the ASQ-3 parent's questionnaire. The advanced neuropsychologist assessment will be done only for patients with CHD with a positive IPA screening.
Performance (negative predictive value) of the IPA screening for NDD on the NDD high risk population | 4 months (to obtain the neurophysiologist assessment)
  This will be evaluated by comparing the results of the IPA screening (using both HAS scale and ASQ-3 parent's questionnaire) with results of the advanced neuropsychologist assessment. A positive IPA screening is defined by a NDD alert using the HAS scale and/or the ASQ-3 parent's questionnaire. The advanced neuropsychologist assessment will be done only for patients with CHD with a positive IPA screening.
Prevalence of NDD in the high risk population | 18 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - University Hospitial of Montpellier, Montpellier
  - Institut Marin Saint-Pierre, Palavas-les-Flots
  - CHU Bordeaux Haut-Lévêque, Pessac